CLINICAL TRIAL: NCT02214550
Title: Deciphering the Hormonal and Nociceptive Mechanisms Underlying Bladder Pain
Brief Title: Chronic Pain Risk Associated With Menstrual Period Pain
Acronym: CRAMPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank Tu, Division Director, Gynecological Pain and Minimally Invasive Surgery, Department of Obstetrics and Gynecology, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EH13-094; 1R01DK100368-01 (NIH)
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Cystitis, Interstitial; Dysmenorrhea; Migraine Disorders; Pelvic Pain; Endometriosis; Visceral Pain; Chronic Pain
Keywords: Cystitis, Interstitial; Dysmenorrhea; Migraine Disorders; Cross Organ Sensitization; Pelvic Pain; Endometriosis; Contraceptives, Oral; Birth Control Pills; Painful Bladder Syndrome; Visceral Pain; Chronic Pain
MeSH Terms: conditions — Cystitis, Interstitial; Dysmenorrhea; Migraine Disorders; Pelvic Pain; Endometriosis; Visceral Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- D+COS-no OC (No Intervention): Ten participants in the Dysmenorrhea + COS group will not receive an OC intervention. Monthly questionnaires will be completed for 1 yr. QST will be repeated at 6 months and 12 months. A yearly follow-up questionnaire will be completed for 5 years.
- D+COS-cyclic microgestin 1/20 (Active Comparator): 26 participants in the Dysmenorrhea + COS group will receive cyclic OC. Monthly questionnaires will be completed for 1 yr. QST will be repeated at 6 months and 12 months. A yearly follow-up questionnaire will be completed for 5 years.
  Interventions: Drug: cyclic microgestin 1/20
- D+COS-continuous microgestin 1/20 (Active Comparator): 26 participants in the Dysmenorrhea + COS group will receive continuous OC. Monthly questionnaires will be completed for 1 yr. QST will be repeated at 6 months and 12 months. A yearly follow-up questionnaire will be completed for 5 years.
  Interventions: Drug: continuous microgestin 1/20
- PBS-continuous microgestin 1/20 (Active Comparator): 26 participants in the Painful Bladder Syndrome group will receive continuous OC. Monthly questionnaires will be completed for 1 yr. QST will be repeated at 6 months and 12 months. A yearly follow-up questionnaire will be completed for 5 years.
  Interventions: Drug: continuous microgestin 1/20
- No Intervention: Pain Discovery Aim (No Intervention): 255 Reproductive-age women (18-45) will be identified and divided into 5 groups
  Healthy Controls Chronic Pain (Positive Controls) Dysmenorrhea (D) Dysmenorrhea with Cross Organ Sensitization (D+COS) Painful bladder syndrome (PBS)/interstitial cystitis (IC) After a screening, dysmenorrhea with COS and PBS participants will be compared with controls. Daily Diaries will be completed for 1-3 months. During the luteal phase of the participants' menstrual cycle or a predetermined time, participants will complete aim #1 testing consisting of a battery of questionnaires, bladder sensitivity testing, quantitative sensory testing (QST), a blood draw and EEG testing. All participants will also complete a yearly follow-up questionnaire for 5 years.

INTERVENTIONS:
Drug: cyclic microgestin 1/20 — Cyclic OC Use - Participants will ingest pills containing active hormones for 21 days followed by 7 days of no pills, and then the cycle will repeat
  Other Names: loestrin 1/20
  Arms: D+COS-cyclic microgestin 1/20
Drug: continuous microgestin 1/20 — Continuous OC use - Pills containing hormones will be taken every day for 1 year
  Other Names: loestrin 1/20
  Arms: D+COS-continuous microgestin 1/20; PBS-continuous microgestin 1/20

SUMMARY:
The purpose of this study is to determine if some women with dysmenorrhea (painful periods) are at higher future risk of developing chronic pelvic pain (CPP) and if oral contraceptives (OC) can be used to reverse this chronic pain risk.

Investigators will examine whether dysmenorrhea produces CPP via repetitive cross organ sensitization (COS) episodes. The use of cyclical OCs to eliminate dysmenorrhea is expected to reduce COS and decrease the risk of developing CPP.

DETAILED DESCRIPTION:
Endometrial shedding during the menstrual cycle elicits profound changes in neuronal activity and cytokine concentrations producing moderate to severe pelvic pain in more than 20% of reproductive-age women. One out of every five of those women in turn will develop chronic pelvic pain (CPP), yet women without dysmenorrhea rarely report CPP. CPP disorders such as irritable bowel syndrome (IBS) and painful bladder syndrome (PBS) can cause severe, unrelenting pain due to a lack of effective treatments.

This study consists of 2 aims.

Aim #1: To determine if dysmenorrhea with concomitant bladder pain sensitivity exhibits neurophysiological features consistent with established CPP. Women with chronic pain or dysmenorrhea without COS will be used as controls. Quantitative sensory testing (QST) and a noninvasive bladder pain test that investigators validated previously be used to determine whether impairments in descending inhibition and pelvic sensitivity are responsible for vulnerability to COS in women with dysmenorrhea. EEG will be recorded to look for differences in brain activity in response to sensory stimulation between participants cohorts.

Aim #2: To differentiate the individual contributions of circulating sex hormones and repeated sensitizing events (painful menses) on descending and peripheral mechanisms of bladder pain. The same QST/bladder pain measures studied in Aim #1 will be retested within the dysmenorrhea+COS group following a one-year randomized trial of cyclical OCs vs. continuous OCs vs. no treatment. An observational arm of PBS participants will receive continuous OCs and serve as controls.

ELIGIBILITY:
Inclusion Criteria:

All

* Reproductive age women (18-45)

For dysmenorrhea and D+COS group only:

* Participants must have had regular (22-45 day) menstrual cycles over at least a two month period preceding testing

Exclusion Criteria:

All

* presence of active pelvic or abdominal malignancies (primary or metastatic)
* active genitourinary infection in the last four weeks
* unable to read or comprehend the informed consent in English
* unwilling to undergo pelvic examination/testing
* presence of hypertension or risk for developing hypertension, and

For dysmenorrhea and D+COS group only:

* absence of regular menses (including current pregnancy, recent pregnancy, or active breast feeding) unwilling to take either cyclic or combined OCs
* unwilling to withdraw from OCs for two months prior to the sensory testing study visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 353 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tu, MD, MPH, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu FF, Epstein AE, Pozolo KE, Sexton DL, Melnyk AI, Hellman KM. A noninvasive bladder sensory test supports a role for dysmenorrhea increasing bladder noxious mechanosensitivity. Clin J Pain. 2013 Oct;29(10):883-90. doi: 10.1097/AJP.0b013e31827a71a3. PMID 23370073
- [Background] Tu FF, Fitzgerald CM, Kuiken T, Farrell T, Norman Harden R. Vaginal pressure-pain thresholds: initial validation and reliability assessment in healthy women. Clin J Pain. 2008 Jan;24(1):45-50. doi: 10.1097/AJP.0b013e318156db13. PMID 18180636
- [Background] Zondervan KT, Yudkin PL, Vessey MP, Jenkinson CP, Dawes MG, Barlow DH, Kennedy SH. Chronic pelvic pain in the community--symptoms, investigations, and diagnoses. Am J Obstet Gynecol. 2001 May;184(6):1149-55. doi: 10.1067/mob.2001.112904. PMID 11349181
- [Background] Westling AM, Tu FF, Griffith JW, Hellman KM. The association of dysmenorrhea with noncyclic pelvic pain accounting for psychological factors. Am J Obstet Gynecol. 2013 Nov;209(5):422.e1-422.e10. doi: 10.1016/j.ajog.2013.08.020. Epub 2013 Aug 22. PMID 23973396
- [Background] Brotzner CP, Klimesch W, Doppelmayr M, Zauner A, Kerschbaum HH. Resting state alpha frequency is associated with menstrual cycle phase, estradiol and use of oral contraceptives. Brain Res. 2014 Aug 19;1577(100):36-44. doi: 10.1016/j.brainres.2014.06.034. Epub 2014 Jul 7. PMID 25010817
- [Derived] Kmiecik MJ, Tu FF, Clauw DJ, Hellman KM. Multimodal hypersensitivity derived from quantitative sensory testing predicts pelvic pain outcome: an observational cohort study. Pain. 2023 Sep 1;164(9):2070-2083. doi: 10.1097/j.pain.0000000000002909. Epub 2023 Apr 27. PMID 37226937

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were drawn from a separate cross-sectional, observational study that included women who mostly had moderate-to-severe dysmenorrhea, but also included some healthy controls, and patients with other chronic pain conditions who served as positive controls for that study. Those with D+COS and PBS in the four intervention arms first participated in the strictly observational study, yielding all baseline data. The Intervention arm participants are NOT included in the "no intervention' arms.
Groups:
- D+COS-no OC: 10 participants in the Dysmenorrhea + COS group will not receive an OC intervention. Monthly questionnaires will be completed for 1 yr. QST will be repeated at 6 months and 12 months. A yearly follow-up questionnaire will be completed for 5 years.
- No Intervention: Healthy Controls: Healthy control cases will have average pain ≤ 3/10 with menses or with withdrawal uterine bleeding from cyclical OCs and b) < 2 migraines per year will be recruiting preferentially.
- No Intervention Chronic Pain (Positive Controls): Chronic Pain (Positive Controls) will have a diagnosed, documented (reviewed by PI) chronic pain disorder greater than six months' duration, which has required at least 2 different prescription treatments and/or surgical management. They must report an average pain of at least 5/10 in the last month. We will accept participants with any type of chronic pain (except for individuals with bilateral knee and hand pain) but anticipate many of our chronic pain participants to suffer from fibromyalgia, lower back pain, and chronic pelvic pain (including irritable bowel syndrome).
- No Intervention: Dysmenorrhea (D): Dysmenorrhea cases will have: a) average menstrual pain ≥ 5/10 (0=no pain and 10=the worst imaginable pain) with menses or withdrawal uterine bleeding from cyclic OCs without painkillers, b) menstrual pain in the region between the umbilicus and the perineum, above the level of the inguinal ligament and c) indication the participant has attempted to resolve pain by medical means (including NSAIDs and/or OCs). Dysmenorrhea ONLY cases will have <16 bladder pain on a 0-100 visual analogue scale (VAS) during either first sensation or first urge at assessment visit #1.
- No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS): will meet criteria for Dysmenorrhea cases, with >15 bladder pain on a 0-100 visual analogue scale (VAS) during either first sensation or first urge at assessment visit #1.
- No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC): Diagnosis of PBS participants will be confirmed by medical records indicating chronic (>3 months) pelvic pain (average intensity ≥ 3/10), pressure, or discomfort related to the bladder accompanied by at least one other urinary symptom such as persistent urge to void or frequency.34 PBS participants will also have records review to confirm the exclusion of other conditions by clinical examination or cystoscopy if necessary. PBS participants can have other chronic pain conditions.
Period: Overall Study
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20 | No Intervention: Healthy Controls | No Intervention Chronic Pain (Positive Controls) | No Intervention: Dysmenorrhea (D) | No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS) | No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC)
Started | 6 | 4 | 8 | 15 | 45 | 39 | 187 | 35 | 14
Baseline | 6 | 4 | 8 | 14 | 37 | 31 | 102 | 34 | 10
Month 6 | 6 | 4 | 5 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 4 | 5 | 6 | 37 | 31 | 102 | 34 | 10
Not Completed | 0 | 0 | 3 | 9 | 8 | 8 | 85 | 1 | 4

BASELINE CHARACTERISTICS:
Population: For PBS-continuous microgestin 1/20, one of the 15 participants who signed consent and came for a screening visit, changed her mind about taking microgestin and did not come for a baseline visit, so the final sample size for that subgroup is n=14
Groups:
- No Intervention: Healthy Controls: Healthy control cases will have average pain ≤ 3/10 with menses or with withdrawal uterine bleeding from cyclical OCs and b) < 2 migraines per year will be recruited preferentially.
- Total: Total of all reporting groups
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20 | No Intervention: Healthy Controls | No Intervention Chronic Pain (Positive Controls) | No Intervention: Dysmenorrhea (D) | No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS) | No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC) | Total
Number analyzed (Participants) | 6 | 4 | 8 | 15 | 37 | 31 | 102 | 34 | 10 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.5) | 20.00 (1.41) | 22.2 (4.06) | 30.4 (5.93) | 23.9 (7.1) | 27.5 (6.2) | 24.1 (6.7) | 24.7 (6.5) | 26.8 (5.5) | 26.1 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 8 | 15 | 37 | 31 | 102 | 34 | 10 | 247
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 3 | 29 | 15 | 7 | 0 | 55
  Not Hispanic or Latino | 5 | 4 | 8 | 15 | 34 | 2 | 87 | 27 | 10 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 3 | 0 | 2 | 0 | 9 | 0 | 15 | 7 | 0 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3 | 3 | 2 | 21 | 6 | 0 | 38
  White | 2 | 4 | 3 | 12 | 21 | 28 | 53 | 20 | 8 | 151
  More than one race | 1 | 0 | 0 | 0 | 2 | 1 | 13 | 1 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bladder Pain Sensitivity [Mean (Standard Deviation); unit: Visual Analog Scale] — Visual Analog Scale is a 0 through 100 scale with 0 being no pain and 100 worst pain imaginable.
  Results from the visual analog scale (VAS) of the bladder filling test will be compared to determine if participants in each of the treatment groups had a reduction in pain. Bladder pain ratings at first urge will be used at the outcome measure. Population: Participant did not report a pain rating for first urge during the bladder test.
  Visual Analog Scale
    number analyzed (Participants) | 6 | 4 | 8 | 14 | 37 | 31 | 102 | 33 | 10 | 245
    (all) | 38.2 (13.5) | 37.0 (10.7) | 41.2 (16.9) | 47.9 (12.9) | 2.2 (2.8) | 17.3 (17.3) | 4.1 (4.2) | 33 (13.9) | 49.0 (26.4) | 43.0 (14.0)
Quantitative Sensory Testing (QST) parameters regarding pelvic hyperalgesia [Mean (Standard Deviation); unit: Newtons] — Amount of pressure applied to the pelvic floor in newtons (0-30) before the first threshold for pain. Population: Malfunctioning digital algometer or pelvic pain testing was too painful for participants to complete testing.
  Newtons
    number analyzed (Participants) | 5 | 4 | 8 | 14 | 37 | 31 | 102 | 34 | 10 | 245
    (all) | 5.95 (3.96) | 9.38 (6.56) | 13.8 (11.9) | 8.21 (6.04) | 11.6 (6.4) | 6.9 (4.5) | 8.9 (5.6) | 7.2 (5.2) | 6.9 (3.2) | 9.43 (7.92)

OUTCOME MEASURES:

1. Primary Outcome: Change in Participant Bladder Pain Sensitivity From Baseline.
Description: Score on a scale. Specifically, we used a Visual Analog Scale- 0 through 100 scale with 0 being no pain and 100 worst pain imaginable. Results from the visual analog scale (VAS) of the bladder filling test at the initial, 6 month and 12 month visits will be compared to determine if participants in each of the treatment groups had a reduction in pain. Bladder pain ratings at first urge will be used at the outcome measure.
Time Frame: 0 (baseline), 6 month, and 12 month visits
Population: Some participant data were missing due to task error or attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20 | No Intervention: Healthy Controls | No Intervention Chronic Pain (Positive Controls) | No Intervention: Dysmenorrhea (D) | No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS) | No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC)
Number analyzed (Participants) | 6 | 4 | 8 | 14 | 37 | 31 | 102 | 33 | 10
score on a scale
  Baseline | 38.2 (13.5) | 37.0 (10.7) | 41.2 (16.9) | 47.9 (12.9) | 2.2 (2.8) | 17.3 (17.3) | 4.1 (4.2) | 33 (13.9) | 49.0 (26.4)
  Month 6: number analyzed (Participants) | 6 | 4 | 5 | 8 | 0 | 0 | 0 | 0 | 0
  Month 6 | 44.5 (18.5) | 32.0 (21.2) | 18.6 (14.7) | 41.4 (21.6) |  |  |  |  |
  Month 12: number analyzed (Participants) | 6 | 4 | 5 | 6 | 0 | 0 | 0 | 0 | 0
  Month 12 | 47.0 (17.3) | 34.0 (23.5) | 8.6 (10.0) | 38.8 (21.1) |  |  |  |  |
Statistical Analysis 1: Comparison: D+COS-no OC vs D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; A linear mixed-effects model was estimated predicting bladder pain at first urge ratings (0-100 visual analog scale) as a function of time (0, 6, 12 month visits), group, and their interaction. Random intercepts were estimated for each participant. The following three orthogonal contrasts were estimated: 1) OCP vs. No OCP, 2) cyclic vs. continuous microgestin, and 3) PBS-continuous microgestin vs. D+COS-continuous microgestin; Test type: Superiority; p = .02, Mixed Models Analysis — The a priori threshold for statistical significance was .05 and p-values were not adjusted for multiple comparisons given a priori orthogonal contrasts; Slope = -1.96, Standard Error of Mean .69 — Parameter reported indicates time x group interaction (OCP vs. No OCP). PBS participants are included in the OCP group
Statistical Analysis 2: Comparison: D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = -1.4597, Standard Error of Mean 0.8245 — Parameter estimated indicates the time x group (Continuous vs. Cyclic OCP) interaction. PBS participants are included in the continuous OCP group
Statistical Analysis 3: Comparison: D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .023, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 1.9186, Standard Error of Mean 0.8121 — Parameter reported indicates a time x group interaction (D+COS-continuous microgestin vs. PBS-continuous microgestin)

2. Secondary Outcome: Change in Quantitative Sensory Testing (QST) Parameters Regarding Pelvic Hyperalgesia From Baseline
Description: Results from the QST testing performed at initial, 6 month and 12 month visits will be compared to determine if participants in each of the treatment groups had a reduction in sensitivity from baseline. Specifically, measure reported is the pressure pain threshold in newtons observed at the transition from pressure to pain transvaginally at the 12 o'clock position (anteriorly against the bladder). Lower values (pressure) indicate greater sensitivity.
Time Frame: 0 (baseline), 6 months and 12 months
Population: Some participants have missing data due to equipment malfunction or reported pain testing as too painful.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20 | No Intervention: Healthy Controls | No Intervention Chronic Pain (Positive Controls) | No Intervention: Dysmenorrhea (D) | No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS) | No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC)
Number analyzed (Participants) | 5 | 4 | 8 | 14 | 37 | 31 | 102 | 34 | 10
Newtons
  Baseline | 5.95 (3.96) | 9.38 (6.56) | 13.8 (11.9) | 8.21 (6.04) | 11.6 (6.4) | 6.9 (4.5) | 8.9 (5.6) | 7.2 (5.2) | 6.9 (3.2)
  Month 6: number analyzed (Participants) | 5 | 4 | 5 | 6 | 0 | 0 | 0 | 0 | 0
  Month 6 | 5.40 (5.71) | 13.9 (12.9) | 12.3 (10.1) | 3.39 (1.93) |  |  |  |  |
  Month 12: number analyzed (Participants) | 4 | 4 | 5 | 5 | 0 | 0 | 0 | 0 | 0
  Month 12 | 7.36 (8.67) | 7.74 (6.13) | 9.94 (6.80) | 5.59 (1.85) |  |  |  |  |
Statistical Analysis 1: Comparison: D+COS-no OC vs D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; A linear mixed-effects model was estimated predicting pressure pain thresholds (in Newtons of force transvaginally measured anteriorly against the bladder) as a function of time (0, 6, 12 month visits), group, and their interaction. Random intercepts were estimated for each participant. The following three orthogonal contrasts were estimated: 1) OCP vs. No OCP, 2) cyclic vs. continuous microgestin, and 3) PBS-continuous microgestin vs. D+COS-continuous microgestin; Test type: Superiority; p = 0.2315, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 0.3716, Standard Error of Mean 0.3056 — Parameter reported indicates time*group interaction (OCP vs. No OCP). PBS participants are included in the OCP group
Statistical Analysis 2: Comparison: D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = 0.2703, Standard Error of Mean 0.3244 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6341, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = -0.1574, Standard Error of Mean 0.3283 — Parameter estimated indicates the time x group (continuous microgestin: D+COS-vs. PBS) interaction

3. Secondary Outcome: Differences in EEG Recorded Cortical Activity Among Participants
Description: We obtained the peak alpha frequency at the right and left parietal occipital electrodes and averages of the two sides were assessed at Baseline, 6 month, and 12 Month to determine whether differences in resting state brain activity at parieto-occipital electrode sites are affected by oral contraceptives
Time Frame: Baseline, 6 months and 12 months
Population: Some participant data were missing due to attrition, or lack of available equipment on day of study
Measure: Mean (Standard Error); unit: Hertz
Groups:
- D+COS-no OC: Ten participants in the Dysmenorrhea + COS group will not receive an OC intervention. EEG's done at baseline will be repeated at 6 months and 12 months.
- D+COS-cyclic Microgestin 1/20: 26 participants in the Dysmenorrhea + COS group will receive cyclic OC. EEG's done at baseline will be repeated at 6 months and 12 months.
  cyclic microgestin 1/20: Cyclic OC Use - Participants will ingest pills containing active hormones for 21 days followed by 7 days of no pills, and then the cycle will repeat
- D+COS-continuous Microgestin 1/20: 26 participants in the Dysmenorrhea + COS group will receive continuous OC. EEG's done at baseline will be repeated at 6 months and 12 months.
  continuous microgestin 1/20: Continuous OC use - Pills containing hormones will be taken every day for 1 year
- PBS-continuous Microgestin 1/20: 26 participants in the Painful Bladder Syndrome group will receive continuous OC. EEG's done at baseline will be repeated at 6 months and 12 months.
  continuous microgestin 1/20: Continuous OC use - Pills containing hormones will be taken every day for 1 year
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20 | No Intervention: Healthy Controls | No Intervention Chronic Pain (Positive Controls) | No Intervention: Dysmenorrhea (D) | No Intervention: Dysmenorrhea With Cross Organ Sensitization (D+COS) | No Intervention: Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC)
Number analyzed (Participants) | 6 | 4 | 6 | 10 | 31 | 31 | 92 | 29 | 10
Hertz
  Baseline | 10.03 (0.26) | 10.0 (0.59) | 10.05 (0.07) | 10.13 (0.08) | 10.03 (0.06) | 10.15 (0.07) | 10.12 (0.04) | 9.96 (0.06) | 10.0 (0.07)
  Month 6: number analyzed (Participants) | 4 | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 0
  Month 6 | 10.10 (0.24) | 10.01 (0.1) | 10.19 (0.26) | 10.16 (0.18) |  |  |  |  |
  Month 12: number analyzed (Participants) | 3 | 4 | 6 | 4 | 0 | 0 | 0 | 0 | 0
  Month 12 | 9.88 (0.17) | 9.97 (0.94) | 9.75 (0.27) | 10.48 (0.29) |  |  |  |  |
Statistical Analysis 1: Comparison: D+COS-no OC vs D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; A linear mixed-effects model was estimated for parieto-occipital peak alpha (Hz) as a function of time (0, 6, 12 month visits), group, and their interaction. Random intercepts were estimated for each participant. The OCP vs No OCP contrast was estimated here:; Test type: Superiority; p = .393, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = .086, Standard Error of Mean .10 — Parameter reported indicates time x group interaction (OCP vs. No OCP). PBS participants are included in the OCP group
Statistical Analysis 2: Comparison: D+COS-cyclic Microgestin 1/20 vs D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; A linear mixed-effects model was estimated for parieto-occipital peak alpha (Hz) as a function of time (0, 6, 12 month visits), group, and their interaction. Random intercepts were estimated for each participant. The cyclic vs. continuous microgestin contrast was run here; Test type: Superiority; p = 0.941, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = .007, Standard Error of Mean .09 — Parameters reported indicates time x group (Continuous vs. Cyclic OCP) interaction. PBS participants are included in the continuous OCP group
Statistical Analysis 3: Comparison: D+COS-continuous Microgestin 1/20 vs PBS-continuous Microgestin 1/20; A linear mixed-effects model was estimated for parieto-occipital peak alpha (Hz) as a function of time (0, 6, 12 month visits), group, and their interaction. Random intercepts were estimated for each participant. The PBS-continuous microgestin vs. D+COS-continuous microgestin contrast was evaluated here; Test type: Superiority; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Slope = .28, Standard Error of Mean .10 — Parameter reported indicates time x group interaction (D+COS-continuous microgestin vs. PBS-continuous microgestin)

ADVERSE EVENTS:
Time Frame: Surveys of adverse events were collected monthly over 1 Year
Description: We used a survey with prespecified questions. Please note, all-cause mortality or serious & other AEs were not monitored in the "no intervention arms". In the intervention arms, no formal query for mortality or serious AE was done, but we did monitor for them. For nonserious AEs, we report the frequency of ever reporting any queried event over the entire period. Participants varied in total AE form completion. Participants in the "D+COS-no OC" group did not receive AE questionnaires.
Arm/Group | D+COS-no OC | D+COS-cyclic Microgestin 1/20 | D+COS-continuous Microgestin 1/20 | PBS-continuous Microgestin 1/20
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/0 | 4/4 | 8/8 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D+COS-no OC (N=0) | D+COS-cyclic Microgestin 1/20 (N=4) | D+COS-continuous Microgestin 1/20 (N=8) | PBS-continuous Microgestin 1/20 (N=6)
Nausea (Nervous system disorders) | 0 | 4 | 8 | 6
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Spotting (between periods) (Reproductive system and breast disorders) | 0 | 4 | 8 | 6
Breast Tenderness (Reproductive system and breast disorders) | 0 | 3 | 6 | 6
Weight Gain (Metabolism and nutrition disorders) | 0 | 4 | 7 | 5
Headache (Nervous system disorders) | 0 | 4 | 7 | 6
Depressed, sad a lot (Psychiatric disorders) | 0 | 4 | 6 | 6
Irritable (Psychiatric disorders) | 0 | 4 | 7 | 6
Darkening of the skin or face (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Decreased sex drive (Reproductive system and breast disorders) | 0 | 3 | 4 | 3
Changes in vision (Eye disorders) | 0 | 3 | 3 | 1

LIMITATIONS AND CAVEATS:
Small sample size due to higher than expected refusal of participants with DYSB to randomize to an OCP limits generalizability. As noted above, nonserious adverse events are reported as the frequency of ever reporting an event on a form, of any intensity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02214550/Prot_SAP_000.pdf